CLINICAL TRIAL: NCT02480101
Title: Reactogenicity, Safety and Immunogenicity of a Live Monovalent A/17/Anhui/2013/61 (H7N9) Influenza Vaccine
Brief Title: Reactogenicity, Safety and Immunogenicity of a LAIV H7N9 Influenza Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Research Institute of Influenza, Russia (Other)
Collaborators: World Health Organization (Other); Institute of Experimental Medicine, Russia (Other)
Responsible Party: Principal Investigator, Oleg Kiselev, Director, Research Institute of Influenza, Russia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LAIV-H7N9-01
Record Dates: First submitted 2015-06-16; First posted 2015-06-24 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-06

CONDITIONS: Influenza
Keywords: influenza vaccine pandemic
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- H7N9 LAIV (Active Comparator): H7N9 live influenza vaccine
  Interventions: Biological: H7N9 live influenza vaccine
- Placebo (Placebo Comparator): Lyophilized purified allantoic fluid of chicken embryos with stabilizers
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: H7N9 live influenza vaccine — H7N9 live influenza vaccine
  Other Names: LAIV H7N9
  Arms: H7N9 LAIV
Biological: Placebo — Lyophilized purified allantoic fluid of chicken embryos with stabilizers
  Arms: Placebo

SUMMARY:
This is a single centre phase I, double-blind placebo-controlled study to assess reactogenicity, safety and immunogenicity of a live monovalent A/17/Anhui/2013/61 (H7N9) influenza vaccine in healthy male and female adults, 18 through 49 years of age .

ELIGIBILITY:
Inclusion Criteria:

* Legal male or female adult 18 through 49 years of age at the enrollment visit.
* Literate and willing to provide written informed consent.
* A signed informed consent.
* Free of obvious health problems, as established by the medical history and screening evaluations, including physical examination.
* Capable and willing to complete diary cards and willing to return for all follow-up visits
* Willing to comply with the rules of the isolation unit (including willing and able to take oseltamivir influenza antiviral medication, should that be recommended by a study physician).
* For females, willing to take reliable birth control measures through day 56.

Exclusion Criteria:

* Participation in another clinical trial involving any therapy within the previous three months or planned enrollment in such a trial during the period of this study.
* Receipt of any non-study vaccine within four weeks prior to enrollment or refusal to postpone receipt of such vaccines until four weeks after study completion.
* Practice of nasal irrigation on a regular basis within the past six months or has engaged in nasal irrigation within two weeks prior to enrollment.
* Recent history of frequent nose bleeds (more than 5 within the past year).
* Clinically relevant abnormal paranasal anatomy.
* Recent history (within the past month) of rhino or sinus surgery, or surgery for any traumatic injury of the nose.
* Current or recent (within two weeks of enrollment) acute respiratory illness with or without fever.
* Other acute illness at the time of study enrollment.
* Receipt of immune globulin or other blood products within three months prior to study enrollment or planned receipt of such products during the period of subject participation in the study.
* Chronic administration (defined as more than 14 consecutively-prescribed days) of immunosuppressants or other immune-modulating therapy within six months prior to study enrollment (for corticosteroids, this means prednisone or equivalent, 0.5 mg per kg per day; topical steroids are allowed, exclusive of nasal.)
* Participation in any previous trial of any H7 or H5 containing influenza vaccine.
* History of bronchial asthma.
* Hypersensitivity and allergy reactions after previous administration of any vaccine.
* History of wheezing after past receipt of any live influenza vaccine.
* Other AE following immunization (body temperature more than 40°C, collapse, non-febrile seizures, anaphylaxis), at least possibly related to previous receipt of any vaccine (not only influenza).
* Suspected or known hypersensitivity to any of the study vaccine components, including chicken or egg protein.
* Seasonal (autumnal) hypersensitivity to the natural environment.
* Acute or chronic clinically significant pulmonary, cardiovascular, hepatic, metabolic, neurologic, psychiatric or renal functional abnormality, as determined by medical history, physical examination or clinical laboratory screening tests, which in the opinion of the investigator, might interfere with the study objectives. Subjects with physical examination findings or clinical laboratory screening results which would be graded 2 or higher on the AE severity grading scale will be excluded from entry into the study and will be excluded from receipt of dose two of study vaccine or placebo.
* History of leukemia or any other blood or solid organ cancer.
* History of thrombocytopenic purpura or known bleeding disorder.
* History of seizures.
* Known or suspected immunosuppressive or immunodeficient condition of any kind, including HIV infection.
* Known chronic HBV or HCV infection.
* Known tuberculosis infection or evidence of previous tuberculosis exposure.
* History of chronic alcohol abuse and/or illegal drug use.
* Claustrophobia or sociophobia.
* Pregnancy or lactation (a negative pregnancy test will be required before administration of study vaccine or placebo for all women of childbearing potential).
* Any condition that, in the opinion of the investigator, would increase the health risk to the subject if he/she participates in the study or would interfere with the evaluation of the study objectives.
* Allergic, including anaphylactic, reactions to the introduction of any vaccines in the subject's medical history (not only flu vaccine).

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2014-10; Primary Completion 2014-12 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Immediate reactions | 2 hours
  Immediate reactions occurring within two hours of administration of any dose, measured as observed by study staff or reported by the subject to study staff
Solicited adverse events | Greater than two hours after administration of any dose of study vaccine or placebo through 6 days following any dose
  Adverse events commonly associated with intranasal vaccination (solicited local and systemic reactions), measured as observed by study staff or reported by the subject to study staff
Changes from baseline in laboratory findings | Days 3, 6 and 34
  Abnormal laboratory findings from blood and urine specimens
Serious adverse events (SAEs) | 4 weeks of receipt of any dose
  All SAEs during 56 days, as observed by study staff, reported by the subject to study staff, or noted by the subject on a diary card, including abnormal laboratory findings from blood specimens collected on Days 28 (pre-vaccination) and 56

SECONDARY OUTCOMES:
Immune responses | Days 0, 28 and 56
  Immune responses was parameterized as the proportion of subjects with at least a four-fold rise after each dose from baseline or as the mean titer after each dose in any of the following:
  * Serum hemagglutination inhibition (HAI) antibodies
  * Serum neutralizing antibodies
  * Serum immunoglobulin class A (IgA) or immunoglobulin class G (IgG) antibodies measured by enzyme-linked immunosorbent assay (ELISA)
  * Secretory IgA antibodies from the nasal mucosa detected in nasal wick specimens using ELISA
  * Secretory IgA antibodies in saliva specimens using ELISA
Virus shedding | Days 0-6 after each dose
  Virus shedding with virus detected by real-time reverse transcriptase polymerase chain reaction rRTPCR in nasal swabs at any time point (at day of vaccination and daily during hospitalization).
Virus stability | Days 0-6 after each dose
  Virus stability (virus detected and sequenced after inoculation into chicken eggs)

OTHER OUTCOMES:
Cellular immune responses (cytokine and T-cell) | Days 0, 28 and 56
  Cellular immune responses (cytokine and T-cell) was measured using isolated peripheral blood mononuclear cells (PBMCs) tested by flow cytometry and/or enzyme-linked immunosorbent spot (ELISPOT) assay.

CONTACTS AND LOCATIONS:
Overall Officials: Larisa G Rudenko, MD PhD DSc, Study Chair — Institute of Experimental Medicine

REFERENCES:
- [Derived] Rudenko L, Isakova-Sivak I, Naykhin A, Kiseleva I, Stukova M, Erofeeva M, Korenkov D, Matyushenko V, Sparrow E, Kieny MP. H7N9 live attenuated influenza vaccine in healthy adults: a randomised, double-blind, placebo-controlled, phase 1 trial. Lancet Infect Dis. 2016 Mar;16(3):303-10. doi: 10.1016/S1473-3099(15)00378-3. Epub 2015 Dec 8. PMID 26673391